CLINICAL TRIAL: NCT05605405
Title: Prevalence and Associated Factors of Functional Gastrointestinal Disorders Among Children Attending Assuit University Children Hospital
Brief Title: Prevalence and Associated Factors of Functional Gastrointestinal Disorders Among Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahlam Osama, Prevalence and associated factors of functional gastrointestinal disorders among children attending Assuit University Children Hospital, Assiut University
Other Study IDs: PAAFOFGDACAAUCH
Record Dates: First submitted 2021-09-22; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The definition of Functional Gastrointestinal Disorders (FGIDs) has changed over time from the absence of organic disease to a stress-related or psychiatric disorder to a motility disorder, and with Rome III, to a disorder of GI functioning, then Rome iv in 2016 defined FGIDs as : disorders of gut-brain interaction. It is a group of disorders classified by GI symptoms related to any combination of the following: motility disturbance, visceral hypersensitivity,altered mucosal and immune function, altered gut microbiota, and altered central nervous system (CNS) processing. FGIDs are observed in infants and young children worldwide with variable frequency related studies done in variable places around the worled show the following results : the prevalence of FGIDs in Chinese infants and young children is 27.3%.and 40 % in south american infants and 30 % of african infants and 35.1 % of infants presented to tertiary care hospital in Istunbul.Turkey.

DETAILED DESCRIPTION:
The etiology of these disorders remains uncertain and thought to be due to subtle alteration of the normal development or maladaptive behavioral response to a variety of internal or external stimuli .As a group of disorders; FGIDs in young children are a major challenge to the already overstretched pediatric gastroenterology services across the world .Infants and young children with FGIDs visit medical professionals more frequently and experience poor quality of life . In addition, FGIDs in infancy are linked with detrimental repercussions such as maternal depression, poor infant and mother bonding,and poor physical growth .

ELIGIBILITY:
Inclusion Criteria:

* Age group 1 to 18 years old

Exclusion Criteria:

* Age group bwlow 1 year and above 18 years

Having other git problem as :

* GIT bleeding
* H pylori infection
* Cow's milk protein allergy or IBD or any other symptoms suggestive to organic GI disease

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children having functional GI symptoms according Rome IV criteria
Sampling Method: Probability Sample
Enrollment: 269 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of functional gastrointestinal disorders among children attending gastrointerology clinic of Assuit University Children Hospital | 50 weeks
  A number will calculated
The associated factors | 50 weeks
  Demographic and social

IPD SHARING:
Plan to Share IPD: Undecided